CLINICAL TRIAL: NCT01732315
Title: Adolescent Vaccination Reminders Using Email
Brief Title: Adolescent Vaccination Reminder Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Michigan (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-0378
Record Dates: First submitted 2012-10-24; First posted 2012-11-22 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Adolescent Vaccination Status
Keywords: Adolescent vaccination; Immunization rates; Barriers to vaccination; Attitudes; Intentions
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccination Email Reminder (Experimental): This group of parents in the study will receive email notifications about due/overdue vaccines for their adolescents. Vaccination records will be reviewed to identify adolescent patients in both practices who are newly eligible for a vaccine and/or overdue for a vaccine at the start of every other month. Email notifications will then be sent to the parents of these children.
  Interventions: Behavioral: Email Notification
- Usual Care (No Intervention): This group of parents in the study will not receive email notifications about due/overdue vaccines for their adolescents.

INTERVENTIONS:
Behavioral: Email Notification — This study will use a targeted email reminder/recall intervention that addresses specific aspects of adolescent under-immunization.
  Arms: Vaccination Email Reminder

SUMMARY:
This protocol describes a study about vaccination uptake among adolescents. The purpose of the study is to determine whether parents who receive email reminders will be more likely to obtain Tdap (tetanus-diphtheria-acellular pertussis), HPV (human papilloma virus), meningococcal, and influenza vaccines for their adolescent children than parents who do not receive email reminders.

DETAILED DESCRIPTION:
Adolescents are a reservoir population for a variety of vaccine preventable diseases (VPDs). Despite this, adolescent vaccination rates lag substantially behind national goals of 80% coverage for adolescent vaccines set forth by Healthy People 2020. This has been particularly the case for the vaccines most recently recommended for adolescents, such as the HPV (human papilloma virus) and seasonal influenza (flu) vaccines; national coverage levels in 2010 for HPV were 32% (for series completion among females only) and 35% for flu vaccine. Uptake levels for the two other adolescent-targeted vaccines, Tdap and meningococcal conjugate (MCV4) vaccines are currently at 69% and 63%, respectively.

A major barrier to increased adolescent vaccination levels is the lack of parental and provider recognition that an adolescent is due for vaccine doses. For providers, there are the dual challenges of getting adolescents to come in for annual preventive care visits and also minimizing "missed opportunities" for vaccination (i.e. clinical interactions with a patient where a needed vaccine could have been provided but was not). Reminder/recall systems are one mechanism to help address both of these challenges for providers while also informing parents about the need for adolescent vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents (Ages 11-18) have children who attend one of 4 participating pediatric practices,
* Parents are able to read and converse in English,
* Parents have an active email address that is associated with their child's medical record,
* Parents have an adolescent whose medical record can be matched with their MCIR record.

Exclusion Criteria:

* Parent age <18 years,
* Parents have an invalid or non-working parent email address,
* Parents have opted out of email communication,
* Prisoners,
* Decisionally challenged participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3783 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
New immunization doses | New immunizations within 60 days of reminder notification
  To examine the effect of email vaccination reminders, new immunization doses of children of parents who receive email vaccination reminders, versus those who do not receive email reminders during the study period will be determined. New doses are those for any of four adolescent vaccines which are administered following the reminder notification, and are subsequently recorded following reminder notifications.

SECONDARY OUTCOMES:
Waived immunization doses | Waived immunizations within 60 days of reminder notification
  To examine the effect of email vaccination reminders, waived immunization doses of children of parents who receive email vaccination reminders, versus those who do not receive email reminders during the study period will be determined. Waived doses are those for any of four adolescent vaccines for which medical, religious, or philosophical waivers are subsequently recorded following reminder notifications.
Historical immunization doses | Historical immunizations within 60 days of reminder notification
  To examine the effect of email vaccination reminders, historical immunization doses of children of parents who receive email vaccination reminders, versus those who do not receive email reminders during the study period will be determined. Historical doses are those for any of four adolescent vaccines which are administered prior to the reminder notification and are subsequently recorded following reminder notifications.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Dombkowski, DrPH, Principal Investigator — University of Michigan; Amanda Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Dombkowski KJ, Cowan AE, Reeves SL, Foley MR, Dempsey AF. The impacts of email reminder/recall on adolescent influenza vaccination. Vaccine. 2017 May 25;35(23):3089-3095. doi: 10.1016/j.vaccine.2017.04.033. Epub 2017 Apr 25. PMID 28455173